CLINICAL TRIAL: NCT00895167
Title: The Effects of Oral Curcumin on Heme Oxygenase-1 (HO-1) in Healthy Male Subjects
Acronym: CUMAHS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel Doberer (Other)
Responsible Party: Sponsor-Investigator, Daniel Doberer, Subinvestigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT - 2008-004900-30
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Heme Oxygenase; Genetic Polymorphism; Healthy Subjects
MeSH Terms: interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- curcumin (Experimental): every subject receives 12 g of oral curcumin
  Interventions: Dietary Supplement: curcumin

INTERVENTIONS:
Dietary Supplement: curcumin — one oral dose of 12 caplets = 12 g curcumin
  Other Names: Curcumin C3 Complex caplets containing:; 1000 mg curcumin and 5 mg bioperine; Lot. Nr.: #BA 08072227

SUMMARY:
Heme oxygenase 1 (HO-1) serves as a protective gene. Induction of HO-1 has therapeutic potential for several indications. The inducibility of HO-1 by curcumin will be evaluated in this pilot study. Furthermore, the influence of a modulating factor of HO-1 gene activity on the dinucleotide guanosine thymine repeat (GT) length polymorphism in the promotor region will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Male patient aged between 18 and 45 years (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) between 18 and 28 kg/m2 (inclusive) at screening.
* 12-lead ECG without clinically relevant abnormalities at screening.
* Hematology, clinical chemistry, and urinalysis test results not deviating from the normal range to a clinically relevant extent at screening.
* Negative results from urine drug screen at screening.
* Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to the study drug or any excipients of the drug formulation.
* Treatment with another investigational drug within 3 weeks prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs.
* Smoking within the last 3 months prior to screening.
* Previous treatment with any prescribed or OTC medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening.
* Regularly intake of curcumin rich food
* Loss of 250 ml or more of blood within 3 months prior to screening.
* Positive results from the hepatitis serology, except for vaccinated subjects, at screening.
* Positive results from the HIV serology at screening.
* Presumed non-compliance.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The maximal HO-1 mRNA expression and HO-1 protein level in PBMCs | 48 hrs

SECONDARY OUTCOMES:
Increase of plasma bilirubin level | 48 hrs

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- See also: Department of Clinical Pharmacology of the Medical University of Vienna — http://www.meduniwien.ac.at/klpharm/